CLINICAL TRIAL: NCT05725603
Title: Clinical and Anatomical Evaluation of Healing of Lesions of the Subscapular Tendon
Acronym: TENDICICA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A02504-39
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shoulder MRI (Experimental): Shoulder MRI will be performed at least 3 years after shoulder surgery
  Interventions: Other: MRI imaging

INTERVENTIONS:
Other: MRI imaging — Shoulder MRI will be performed at least 3 years after shoulder surgery

SUMMARY:
This study is based on the hypothesis that fatty infiltration postoperative is not or only slightly modified after an atomic repair of lesions of the subscapularis tendon according to a new arthroscopic classification.

DETAILED DESCRIPTION:
After repair of isolated lesions of the subscapularis, it is observed, in nearly half of the cases, a increased fatty infiltration of the subscapularis muscle indicating a probable persistence of the tendon rupture while the Healing failure rate is recognized as moderate (about 15%).

This study is based on the hypothesis that fatty infiltration postoperative is not or only slightly modified after an atomic repair of lesions of the subscapularis tendon according to a new arthroscopic classification.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged ≥ 18 years
* Patient who has undergone surgical repair for a rupture or rotator cuff injury involving the subscapularis tendon between April and September 2016 and between May 2018 and January 2019
* Patient with a lesion of the subscapularis tendon characterized with arthroscopic classification
* Patient who has previously participated in the classification study of subscapularis tendon injuries based on findings arthroscopy conducted only at the Jean Mermoz Hospital

Exclusion Criteria:

* Patient with a contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tendon scarring | 1 day
  Tendon scarring is based on the Sugaya classification from an MRI

SECONDARY OUTCOMES:
Fatty infiltration | 1 day
  The fatty infiltration of the subscapularis muscle is evaluated according to Goutallier's classification

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No